CLINICAL TRIAL: NCT01381172
Title: Evaluation of the Safety and Efficacy of the OPTIMIZER® System in Subjects With Moderate-to-Severe Heart Failure With Ejection Fraction Between 25% and 45%: FIX-HF-5C
Brief Title: Evaluate Safety and Efficacy of the OPTIMIZER® System in Subjects With Moderate-to-Severe Heart Failure: FIX-HF-5C
Acronym: FIX-HF-5C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP OPT2009-009; G030099 (Other: FDA)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: NYHA Class III Heart Failure; NYHA Class IV Heart Failure
Keywords: Heart Failure; Congestive Heart Failure; Chronic heart disease; Cardiac contractility modulation; CCM; CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): The treatment group receives the OPTIMIZER System implant and continues with optimal heart failure medical therapy.
  Interventions: Device: Optimizer System
- Control (Other): The Control group will not receive the OPTIMIZER System and will continue with optimal heart failure medical therapy.
  Interventions: Other: No intervention: Optimal medical therapy

INTERVENTIONS:
Device: Optimizer System — The OPTIMIZER System delivers non-excitatory cardiac contractility modulating (CCM) electrical signals to the heart muscle. Treatment group subjects receive five non-contiguous one-hour periods of CCM signals per day.
  Other Names: CCM therapy
  Arms: Treatment
Other: No intervention: Optimal medical therapy — The control group receives optimal medical therapy only.
  Arms: Control

SUMMARY:
The objective of this investigation is to evaluate the safety and effectiveness of the OPTIMIZER® System in subjects with medically refractory moderate-to-severe heart failure.

DETAILED DESCRIPTION:
The Impulse Dynamics FIX-HF-5C Study is a prospective, multicenter, randomized study to evaluate the safety and efficacy of cardiac contractility modulation (CCM) signals delivered by the implantable OPTIMIZER System in patients with NYHA class III and IV heart failure and an ejection fraction 25-45%. The study will involve the recruitment of 160 subjects at a total of up to 60 sites.

Those subjects who fulfill all inclusion and exclusion criteria based upon baseline test results will be randomly assigned in a 1:1 ratio to either the OPTIMIZER System plus optimal medical therapy (OMT) or to a control group receiving OMT alone. All randomized subjects will be followed for 24 weeks and shall receive the same study related assessments throughout the course of the study. In addition, all subjects will continue to receive OMT for the treatment of their heart failure. Mortality will be reported out to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are 18 years of age or older
2. Subjects who are either male or female. Females of childbearing potential must be using a medically approved method of birth control and must agree to continue to use birth control throughout the study, or must be surgically sterilized (tubal ligation, hysterectomy) or post-menopausal for at least 1 year.
3. Condition

   1. Subjects who have a baseline ejection fraction greater than or equal to 25% and less than or equal to 45% by echocardiography determined by the echocardiography core laboratory.
   2. Subjects who have been treated for heart failure for at least 90 days (including treatment with a β-blocker for at least 90 days unless the subject is intolerant) and are in New York Heart Association functional Class III and IV at the time of enrollment.
   3. Subjects receiving appropriate, stable medical therapy during the 30 days prior to enrollment for treatment of heart failure according to the region- specific guideline recommendations. For patients with EF≤35%, this regimen shall consist of the appropriate doses of diuretics, ACE-inhibitor or angiotensin II receptor blocker and β-blocker. Stable is defined as no more than a 100% increase or 50% decrease in dose.
   4. Subjects who, in the opinion of the Principal Investigator (based on the current guidelines for clinical practice ), have a clinical indication for an implanted cardiac defibrillator (ICD, e.g., EF≤35%) and/or pacemaker, must have an existing device or agree to undergo implantation of such a device unless the patient refuses to undergo the implantation of such device for personal reasons.
   5. Subjects who are willing and able to return for all follow-up visits.

Exclusion Criteria:

1. Subjects whose baseline peak VO2 is <9 or >20 ml O2/min/kg.
2. Subjects who have a potentially correctible cause of heart failure, such as valvular heart disease or congenital heart disease.
3. Subjects who have clinically significant angina pectoris, consisting of angina during daily life (i.e., Canadian Cardiovascular Society Angina score of II or more), an episode of unstable angina within 30 days of enrollment, or angina and/or ECG changes during exercise testing performed during baseline evaluation.
4. Subjects who have been hospitalized for heart failure which required the use of inotropic support within 30 days of enrollment.
5. Subjects who have a clinically significant amount of ambient ectopy, defined as more than 8,900 PVCs per 24 hours on baseline Holter monitoring.
6. Subjects having a PR interval greater than 375 ms.
7. Subjects who have chronic (permanent or persistent) atrial fibrillation or atrial flutter or those cardioverted within 30 days of enrollment.
8. Subjects whose exercise tolerance is limited by a condition other than heart failure (e.g., angina, COPD, peripheral vascular disease, orthopedic or rheumatologic conditions) or who are unable to perform baseline stress testing.
9. Subjects who are scheduled for a CABG or a PTCA procedure, or who have undergone a CABG procedure within 90 days or a PTCA procedure within 30 days of enrollment.
10. Subjects who have a biventricular pacing system, an accepted indication for such a device, or a QRS width of 130ms or greater.
11. Subjects who have had a myocardial infarction within 90 days of enrollment.
12. Subjects who have mechanical tricuspid valve.
13. Subjects who have a prior heart transplant.
14. Subjects on dialysis.
15. Subjects who are participating in another experimental protocol.
16. Subjects who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-01; Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Burkhoff, MD, PhD, Study Director — Impulse Dynamics
Locations (42):
- United States (32):
  - Cardiovascular Consultants, Glendale, Arizona
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - Arizona Heart & Rhythm Center, Phoenix, Arizona
  - Pima Heart, Tucson, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Florida Hospital, Orlando, Florida
  - Florida Hospital - Pepin Heart Institute, Tampa, Florida
  - Advocate Medical Group - Midwest Heart Foundation, Naperville, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Ochsner Clinic, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Detroit Medical Center - Cardiovascular Institute, Detroit, Michigan
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Bryan Heart LGH, Lincoln, Nebraska
  - UMDNJ, Newark, New Jersey
  - Mt. Sinai Medical Center, New York, New York
  - The Lindner Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Guthrie Medical Group, Sayre, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Trinity Clinic, Tyler, Texas
  - Inova Heart & Vascular Institute, Falls Church, Virginia
  - Aurora Health Care, Milwaukee, Wisconsin
- Na Homolce Hospital, Prague, Czechia
- Germany (9):
  - Universitätsmedizin Göttingen, Hanover, Göttingen
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Charité Berlin - Campus Benjamin Franklin, Berlin
  - Charité Campus-Virchow-Klinikum, Berlin
  - ASKLEPIOS Klinik St. Georg, Hamburg
  - UKE - Universitäres Herzzentrum GmbH, Hamburg
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum der Univ. München - Grosshadern, München

REFERENCES:
- [Background] Kadish A, Nademanee K, Volosin K, Krueger S, Neelagaru S, Raval N, Obel O, Weiner S, Wish M, Carson P, Ellenbogen K, Bourge R, Parides M, Chiacchierini RP, Goldsmith R, Goldstein S, Mika Y, Burkhoff D, Abraham WT. A randomized controlled trial evaluating the safety and efficacy of cardiac contractility modulation in advanced heart failure. Am Heart J. 2011 Feb;161(2):329-337.e1-2. doi: 10.1016/j.ahj.2010.10.025. PMID 21315216
- [Background] Abraham WT, Burkhoff D, Nademanee K, Carson P, Bourge R, Ellenbogen KA, Parides M, Kadish A; FIX-HF-5 Investigators and Coordinators. A randomized controlled trial to evaluate the safety and efficacy of cardiac contractility modulation in patients with systolic heart failure: rationale, design, and baseline patient characteristics. Am Heart J. 2008 Oct;156(4):641-648.e1. doi: 10.1016/j.ahj.2008.05.019. PMID 18926146
- [Background] Neelagaru SB, Sanchez JE, Lau SK, Greenberg SM, Raval NY, Worley S, Kalman J, Merliss AD, Krueger S, Wood M, Wish M, Burkhoff D, Nademanee K. Nonexcitatory, cardiac contractility modulation electrical impulses: feasibility study for advanced heart failure in patients with normal QRS duration. Heart Rhythm. 2006 Oct;3(10):1140-7. doi: 10.1016/j.hrthm.2006.06.031. Epub 2006 Jul 8. PMID 17018340
- [Background] Abraham WT, Nademanee K, Volosin K, Krueger S, Neelagaru S, Raval N, Obel O, Weiner S, Wish M, Carson P, Ellenbogen K, Bourge R, Parides M, Chiacchierini RP, Goldsmith R, Goldstein S, Mika Y, Burkhoff D, Kadish A; FIX-HF-5 Investigators and Coordinators. Subgroup analysis of a randomized controlled trial evaluating the safety and efficacy of cardiac contractility modulation in advanced heart failure. J Card Fail. 2011 Sep;17(9):710-7. doi: 10.1016/j.cardfail.2011.05.006. Epub 2011 Jun 22. PMID 21872139
- [Background] Abraham WT, Lindenfeld J, Reddy VY, Hasenfuss G, Kuck KH, Boscardin J, Gibbons R, Burkhoff D; FIX-HF-5C Investigators and Coordinators. A randomized controlled trial to evaluate the safety and efficacy of cardiac contractility modulation in patients with moderately reduced left ventricular ejection fraction and a narrow QRS duration: study rationale and design. J Card Fail. 2015 Jan;21(1):16-23. doi: 10.1016/j.cardfail.2014.09.011. Epub 2014 Oct 5. PMID 25285748
- [Background] Abraham WT, Kuck KH, Goldsmith RL, Lindenfeld J, Reddy VY, Carson PE, Mann DL, Saville B, Parise H, Chan R, Wiegn P, Hastings JL, Kaplan AJ, Edelmann F, Luthje L, Kahwash R, Tomassoni GF, Gutterman DD, Stagg A, Burkhoff D, Hasenfuss G. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Cardiac Contractility Modulation. JACC Heart Fail. 2018 Oct;6(10):874-883. doi: 10.1016/j.jchf.2018.04.010. Epub 2018 May 10. PMID 29754812
- See also: Impulse Dynamics Website — http://www.impulse-dynamics.com/us/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 74 | 86
Completed | 64 | 73
Not Completed | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 74 | 86 | 160
Age, Continuous [Median (Full Range); unit: years] | 61.4 [32 to 85] | 60.0 [28 to 87] | 60.7 [58.5 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 52 | 70 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 15 | 29
  White | 55 | 61 | 116
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 74 | 136
  Czechia | 1 | 3 | 4
  Germany | 11 | 9 | 20
Peak VO2 (ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] — Peak VO2 measures the highest value of oxygen consumption measured during incremental exercise attained during an incremental exercise test, designed to bring the subject to the limit of their exercise tolerance.
  ml/kg/min | 15.36 (2.81) | 15.49 (2.61) | 15.425 (0.141)
Minnesota Living with Heart Failure Questionnaire (MLWHFQ) score [Mean (Standard Deviation); unit: Score on a scale] — Minnesota Living with Heart Failure Questionnaire (MLWHFQ) score. There are 21 questions completed by the participant, with each response on a scale of 0-5. The total score ranges from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
  Score on a scale | 57.35 (23.36) | 56.42 (22.95) | 56.885 (0.28991)
NYHA Class III [Count of Participants; unit: Participants] — Class I: Ordinary physical activity does not cause undue dyspnea or fatigue.
  Class II: Comfortable at rest. Ordinary physical activity results in dyspnea or fatigue.
  Class III: Comfortable at rest. Less than ordinary physical activity results in dyspnea or fatigue.
  Class IV: Symptoms of heart failure may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  Participants | 64 | 78 | 142
NYHA Class IV [Count of Participants; unit: Participants] — Class I: Ordinary physical activity does not cause undue dyspnea or fatigue.
  Class II: Comfortable at rest. Ordinary physical activity results in dyspnea or fatigue.
  Class III: Comfortable at rest. Less than ordinary physical activity results in dyspnea or fatigue.
  Class IV: Symptoms of heart failure may be present even at rest. If any physical activity is undertaken, discomfort is increased.
  Participants | 10 | 8 | 18
6 Minute Hall Walk (meters) [Mean (Standard Deviation); unit: meters] | 324.07 (89.71) | 316.85 (88.37) | 320.46 (0.94045)

OUTCOME MEASURES:

1. Primary Outcome: Peak VO2
Description: Exercise tolerance quantified by peak VO2 measured with cardiopulmonary exercise stress testing (CPX) and evaluated by a blinded core lab.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
ml/kg/min | 15.28 (3.66) | 14.79 (3.54)
Statistical Analysis 1: Comparison: Treatment vs Control; The FIX-HF-5C Study was a study designed to confirm the preliminary evidence reported in the FIX-HF-5 subgroup analysis demonstrating improvement in subjects with LVEF 25-45% and NYHA class III-IV. A Bayesian statistical approach was employed to leverage the data available, particularly the pVO2 results, from the FIX-HF-5 subgroup; Test type: Other — The primary analysis employed a Bayesian repeated measures linear model to estimate group differences in mean pVO2 at 24 weeks from baseline, with 30% borrowing of information (70% down-weighting) from the corresponding treatment group difference observed in the FIX-5 study subgroup. The Bayesian posterior probability would need to be > 0.975 to be considered a positive result with statistical significance; p = 0.975, Bayesian posterior probability — The posterior probability (Pr) that the mean difference in pVO2 (Δ3) between device and control groups is greater than zero must exceed 0.975 to meet the primary effectiveness endpoint

2. Secondary Outcome: Minnesota Living With Heart Failure (MLWHF) Questionnaire
Description: Change in quality of life at 24 weeks compared to baseline, as assessed by the Minnesota Living with Heart Failure (MLWHF) Questionnaire. The MLWHFQ score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of lif
Time Frame: 24 weeks
Population: Randomized subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
score on a scale | 35.26 (24.63) | 47.47 (25.65)

3. Secondary Outcome: Peak VO2 With Respiratory Exchange Ratio (RER)
Description: Peak VO2 with change in respiratory exchange ratio (RER) included as a covariate, as measured by a blinded core lab.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
ml/kg/min | 15.55 (3.51) | 15.25 (3.21)

4. Secondary Outcome: NYHA
Description: Heart failure class, as assessed by the New York Heart Association (NYHA) classification.
Time Frame: 24 weeks
Population: Improvement of 1 NYHA class or more.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
Participants | 57 | 32

5. Secondary Outcome: Peak VO2 With a Peak RER of ≥1.05
Description: Peak VO2 in an analysis that only includes tests with a peak RER of ≥1.05.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
ml/kg/min | 1.13 (0.96) | 1.1 (0.96)

6. Other Pre Specified Outcome: 6 Minute Hall Walk
Description: Distance walked in 6 minutes
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
meters | 324 (90) | 317 (88)

7. Other Pre Specified Outcome: VE/VCO2
Description: VE/VCO2 measured during cardiopulmonary stress testing (CPX) and evaluated by a blinded core lab.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Treatment | Control
Number analyzed (Participants) | 74 | 86
unitless | 15.0 (9.0) | 14.7 (6.0)

ADVERSE EVENTS:
Time Frame: 24 Weeks Study Period
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 1/74 | 4/86
Serious Adverse Events (participants affected / at risk) | 20/74 | 19/86
Other Adverse Events (participants affected / at risk) | 35/74 | 36/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=74) | Control (N=86)
Worsening Heart Failure (Cardiac disorders) | 3 (4) | 7 (8)
Arrhythmia (Cardiac disorders) | 3 (3) | 2 (2)
General Cardiopulmonary (Cardiac disorders) | 3 (4) | 2 (2)
Bleeding (General disorders) | 0 (0) | 1 (1)
Thromboembolism (Cardiac disorders) | 1 (1) | 1 (1)
Local Infection (Infections and infestations) | 1 (1) | 4 (4)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
ICD or Pacemaker System Related (Surgical and medical procedures) | 2 (2) | 0 (0)
OPTIMIZER System Related (Surgical and medical procedures) | 6 (6) | 0 (0)
General Medical (General disorders) | 18 (28) | 17 (29)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=74) | Control (N=86)
Arrhythmias (Cardiac disorders) | 4 (4) | 5 (5)
Bleeding (General disorders) | 2 (2) | 1 (1)
General Cardiopulmonary Event (Cardiac disorders) | 7 (9) | 6 (6)
General Medical (General disorders) | 18 (28) | 17 (29)
ICD or Pacemaker System Related (Surgical and medical procedures) | 2 (2) | 0 (0)
Localized Infection (Infections and infestations) | 5 (5) | 3 (3)
OPTIMIZER System Related (Surgical and medical procedures) | 8 (9) | 0 (0)
Worsening Heart Failure (Cardiac disorders) | 9 (11) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT01381172/Prot_SAP_ICF_000.pdf